CLINICAL TRIAL: NCT06082934
Title: An Open, Prospective, Single-arm Study of Olverembatinib Plus Venetoclax and Dexamethasone in Patients of Newly-diagnosed Ph+ Acute Lymphoblastic Leukemia
Brief Title: Olverembatinib Plus Venetoclax and Dexamethasone for Treatment-naïve Ph+ Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20232082
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2022-11

CONDITIONS: Newly-diagnosed Ph+ Acute Lymphoblastic Leukemia
MeSH Terms: interventions — olverembatinib; venetoclax; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OVD regimen of Olverembatinib plus venetoclax and dexamethasone (Experimental): Olverembatinib: orally every other day at a dose of 40mg Venetoclax: in a daily ramp-up strategy (100 mg d4, 200 mg d5, 400 mg d6-17) Dexamethasone: intravenously 10mg, d1-14, 5mg, d15-28
  Interventions: Drug: Olverembatinib plus venetoclax and dexamethasone

INTERVENTIONS:
Drug: Olverembatinib plus venetoclax and dexamethasone — Olverembatinib: orally every other day at a dose of 40mg Venetoclax: in a daily ramp-up strategy (100 mg d4, 200 mg d5, 400 mg d6-17) Dexamethasone: intravenously 10mg, d1-14, 5mg, d15-28

SUMMARY:
The purpose of this study is to explore the efficacy and safety of the OVD chemotherapy-free regimen (Olverembatinib, venetoclax and dexamethasone) in patients with newly-diagnosed Ph+ALL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

To determine the Complete remission (CR) and complete remission with incomplete hematologic recovery (CRi) rates, the measurable residual disease (MRD) rates, the complete molecular remissions (CMR) rates and the progression-free survival (PFS) of the OVD chemotherapy-free regimen (Olverembatinib, venetoclax and dexamethasone) in patients with newly-diagnosed Ph+ALL.

SECONDARY OBJECTIVES:

To describe the toxicities of the OVD regimen. To assess the quality of life and overall survival of the OVD chemotherapy-free regimen in patients with newly-diagnosed Ph+ALL.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of newly-diagnosed Ph+ acute lymphoblastic leukemia
* Age >= 18
* Adequate hepatic function
* Adequate renal function
* Adequate heart function
* Life expectancy of more than 3 months
* Women of child-bearing potential and men with partners of child-bearing potential must agree to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity from the time of signing the informed consent for through 120 days after the last dose of study medication.
* Women of childbearing potential have negative pregnancy test within 72 hours of initiating study drug dosing.
* Male subjects must agree to use a latex condom during sexual contact with females of childbearing potential even if they have had a successful vasectomy starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* All subjects must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the POMALYST REMS program.

Exclusion Criteria:

* Current or anticipated use of other investigational agents.
* Female patients who are lactating or have a positive serum pregnancy test during the screening period.
* Major surgery within 3 weeks prior to first dose
* Acute active infection requiring systemic antibiotics, antivirals, or antifungals within two weeks prior to first dose
* Known or suspected HIV infection, known HIV seropositivity
* Active hepatitis infection
* Has known chronic obstructive pulmonary disease with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal
* Known gastrointestinal disease or procedure that could interfere with the oral absorption or tolerance, including difficulty swallowing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Complete remission (CR) and complete remission with incomplete hematologic recovery (CRi) rates | Three years
Negative measurable residual disease (MRD) rates | Three years
Complete molecular remissions (CMR) rates | Three years
Progression-free survival (PFS) | Three years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology, Xijing Hospital, Fourth Military Medical University, Xi'an, Shannxi, China